CLINICAL TRIAL: NCT02770287
Title: Clinical Evaluation of the Safety and Efficacy of Using Multi-Polar Radio Frequency and Pulsed Electromagnetic Field Therapy Technologies for the Treatment of the Mon Pubis, Vaginal Introitus and Labia Skin Laxity
Brief Title: Radiofrequency and Pulsed Electromagnetic Field Treatment of Skin Laxity of the Mon Pubis, Labia and Vaginal Introitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS2815
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Masking Description: Independent reviewer to identify the four-month photograph of the mons pubis and labia as compared to the baseline (untreated photo).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venus Freeze Diamond Polar treatment (Experimental): Subjects will receive three treatments with the study device, at four week intervals, followed by a one month follow-up visit after the last treatment.
  Interventions: Device: Venus Freeze Diamond Polar

INTERVENTIONS:
Device: Venus Freeze Diamond Polar — The Venus Freeze Diamond Polar is a non-invasive dermatological treatment system that combines Multi Polar Radiofrequency and Pulsed Magnetic Fields. The radiofrequency energy penetrates the skin and results in tissue heating that has known effect on skin laxity, the magnetic field that is simultaneously induces increases fibroblast collagen production through non thermal mechanism and contributes to the clinical effect of skin laxity improvement. Only the Diamond Polar applicator will be used in this study for the treatment of the Mons pubis, vaginal introitus and Labia. Minor modification to the hand-piece for operator and/or patient comfort may occur mid-study, however no change in range of energy modality or amount of energy delivered will occur at any point during the study.

SUMMARY:
The study will confirm that the Freeze Diamond polar applicator is safe for treating the Mons pubis and Labia, and will result in improvement in general skin appearance including an improvement in skin irregularities and skin laxity.

DETAILED DESCRIPTION:
This is a single-center, open-label, prospective study. Ten (10) subjects that meet the inclusion criteria will be enrolled from the site's pool of patients. Subjects should be a female at the age of 25-65, and have a suitable treatment area (e.g. skin irregularities and/or unwanted skin laxity in the Mons pubis, Introitus and/or Labia area).

Subjects will receive three treatments with the study device, at four week intervals, followed by one month follow-up visits after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female between the ages of 25 and 65.
2. Able to read, understand and voluntarily provide written Informed Consent;
3. Able and willing to comply with the treatment/follow-up schedule and requirements;
4. Fitzpatrick skin type I-VI.
5. Sexual activity (vaginal intercourse once per month) in a monogamous relationship.
6. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment, and have a negative Urine Pregnancy test at baseline.
7. Women requesting aesthetic benefit to the vaginal mons, introitus and labia.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the course of study. A urine pregnancy test will be given to women of childbearing potential and performed during initial visit.
2. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Having a permanent implant in the treated area.
4. Prior use of retinoids in treated area within 2 weeks of initial treatment or during the course of the study.
5. Use of oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study.
6. Patient on systemic corticosteroid therapy 6 months prior to and throughout the course of the study.
7. Prior skin treatment with laser in treated area within 6 months of initial treatment or during the course of the study.
8. Prior use of collagen, fat injections and /or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 4-6 weeks of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants.
9. Prior ablative resurfacing procedure in treated area with laser or other devices within 12 months of initial treatment or during the course of the study.
10. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
11. History of keloid formation or poor wound healing in a previously injured skin area.
12. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
13. Open laceration or abrasion of any sort on the area to be treated.
14. Active sexually transmitted disease (e.g. genital Herpes Simplex, condylomata) or vaginosis; any tissue biopsy will be deferred or delayed to a later time point until the infection is resolved.
15. Chronic vulvar pain or vulvar dystrophy.
16. History of immunosuppression/immune deficiency disorders (including human immunodeficiency virus infection or acquired immune deficiency syndrome) or use of immunosuppressive medications.
17. Having any form of active cancer at the time of enrollment and during the course of the study.
18. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the treatment, or healing process.
19. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria.
20. Tattoos in the treatment area.
21. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse.
22. Having any stage 3-4 cystocele, rectocele, enterocele paravaginal defect or major pelvic organ prolapse beyond the hymenal ring.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Reiz, Study Director — Venus Concept
Locations (1):
- Revive Wellness Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center, baseline-controlled, open-label study. First subject enrolled March 26, 2016 and last subject completed the study on June 28, 2016.
Groups:
- Treatment Group: Subjects will receive three treatments with the study device, at four week intervals, followed by a one month follow-up visit after the last treatment.
  Venus Freeze Diamond Polar: The Venus Freeze Diamond Polar is a non-invasive dermatological treatment system combines Multi Polar Radiofrequency and Pulsed Magnetic Fields. The radiofrequency energy penetrates the skin and results in tissue heating that has known effect on skin laxity, the magnetic field that is simultaneously induces increases fibroblast collagen production through non thermal mechanism and contributes to the clinical effect of skin laxity improvement. Only the Diamond Polar applicator will be used in this study for the treatment of the Mons pubis, vaginal introitus and Labia. Minor modification to the hand-piece for operator and/or patient comfort may occur mid-study, however no change in range of energy modality or amount of energy delivered will occur at any point during the study.
Period: Overall Study
Arm/Group | Treatment Group
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Venus Freeze Diamond Polar: Subjects will receive three treatments with the study device, at four week intervals, followed by a one month follow-up visit after the last treatment.
  Venus Freeze Diamond Polar: The Venus Freeze Diamond Polar is a non-invasive dermatological treatment system combines Multi Polar Radiofrequency and Pulsed Magnetic Fields. The radiofrequency energy penetrates the skin and results in tissue heating that has known effect on skin laxity, the magnetic field that is simultaneously induces increases fibroblast collagen production through non thermal mechanism and contributes to the clinical effect of skin laxity improvement. Only the Diamond Polar applicator will be used in this study for the treatment of the Mons pubis, vaginal introitus and Labia. Minor modification to the hand-piece for operator and/or patient comfort may occur mid-study, however no change in range of energy modality or amount of energy delivered will occur at any point during the study.
Arm/Group | Venus Freeze Diamond Polar
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Baseline photograph of treatment area [Number; unit: participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: General Skin Appearance of Mons Pubis and Labia
Description: Improvement in general skin appearance at follow-up visit 3 as compared to baseline as assessed by independent blinded evaluator by photographic assessment, utilizing the Global Aesthetic Improvement Scale (GAIS) where 3 = very much improved, 2 = much improved, 1 = improved, 0 = no change, -1 = worse, -2 = much worse and -3 = very much worse where higher scores indicate a better outcome.
Time Frame: Baseline - Day 1, Follow-up visit - Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | Venus Freeze Diamond Polar
Number analyzed (Participants) | 8
Participants
  GAIS Very Much Improved | 3
  GAIS Much Improved | 4
  GAIS Improved | 1

2. Secondary Outcome: Visual Analogue Scale (VAS)
Description: The subject records their measure of discomfort and pain associated with all treatments of the labia as a vertical line drawn on a 100 mm horizontal line on which the discomfort and pain intensity is represented by a point between the extremes of "no pain at all" (a value of 0 mm) and "worst pain imaginable (a value of 100 mm).
Time Frame: Treatment 1 - Day 1, Treatment 2 - Day 29, Treatment 3 - Day 57
Population: Subjects reported 26 VAS scores for treatment 1, treatment 2 and treatment 3 of the labia
Measure: Mean (Full Range); unit: score on a scale
Groups:
- VAS - Labia Treatment: Subjects recorded their assessment of pain on the 10cm Visual Analogue Scale (VAS) after each treatment.
Arm/Group | VAS - Labia Treatment
Number analyzed (Participants) | 26
score on a scale
  Treatment 1 | 1.6 [0.1 to 7.3]
  Treatment 2 | 1.7 [0.2 to 7.9]
  Treatment 3 | 1.9 [0.1 to 6.6]

3. Secondary Outcome: Visual Analog Scale (VAS)
Description: The subject records their measure of discomfort and pain associated with all treatments of the mons pubis as a vertical line drawn on a 100 mm horizontal line on which the discomfort and pain intensity is represented by a point between the extremes of "no pain at all" (a value of 0 mm) and "worst pain imaginable (a value of 100 mm).
Time Frame: Treatment 1 - Day 1, Treatment 2 - Day 29, Treatment 3 - Day 57
Population: Subjects reported 26 VAS scores for treatment 1, treatment 2 and treatment 3 of the mons pubis
Measure: Mean (Full Range); unit: score on a scale
Groups:
- VAS - Mons Pubis Treatment: Subjects re
Arm/Group | VAS - Mons Pubis Treatment
Number analyzed (Participants) | 26
score on a scale
  Treatment 1 | 1.2 [0.1 to 3.8]
  Treatment 2 | 0.9 [0.1 to 2.8]
  Treatment 3 | 1.2 [0.1 to 3.5]

4. Secondary Outcome: Vaginal pH
Description: Vaginal pH was obtained at each study visit. The pH is a numeric value from 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 is neutral, lower values are more acidic (value of 0) and higher values more alkaline (value of 14). A healthly vaginal pH has a value of 3.8 to 4.5.
Time Frame: Treatment 1 - Day 1, Treatment 2 - Day 29, Treatment 3 - Day 57, Follow-up visit - Day 85
Population: Vaginal pH was obtained for 11 subjects at the treatment 1 visit, 9 subjects for the treatment 2 visit, 8 subjects for the treatment 3 visit and only 5 subjects at the follow up visit. No baseline vaginal pH's were obtained.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Vaginal pH: The vaginal pH was obtained from all subjects at each visit.
Arm/Group | Vaginal pH
Number analyzed (Participants) | 11
score on a scale
  Treatment 1 | 4.5 [3.9 to 4.8]
  Treatment 2: number analyzed (Participants) | 9
  Treatment 2 | 4.3 [3.9 to 4.5]
  Treatment 3: number analyzed (Participants) | 8
  Treatment 3 | 4.4 [4.2 to 4.5]
  Follow up Visit: number analyzed (Participants) | 5
  Follow up Visit | 4.3 [4.1 to 4.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months and 2 days.
Arm/Group | Venus Freeze Diamond Polar
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venus Freeze Diamond Polar (N=11)
Vaginal canal pain (Reproductive system and breast disorders) | 1 (1)
Pain, biopsy site (Skin and subcutaneous tissue disorders) | 2 (2)
Achy cramps, contractions (Reproductive system and breast disorders) | 1 (1)
Blistering inside vaginal canal (Reproductive system and breast disorders) | 1 (1)
Feeling of 'blistering' inside vaginal canal (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02770287/Prot_SAP_000.pdf